CLINICAL TRIAL: NCT02534532
Title: Atrial Fibrillation Screening With a Smartphone Device and iECG Application
Acronym: AFScreenCol
Status: Withdrawn | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18250
Record Dates: First submitted 2015-08-19; First posted 2015-08-27 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation screening
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Females and males ≥65 years old, attending to the primary care centers, located in three different major cities in Colombia, that are willing to participate in the study, and do not present any exclusion criteria
  Interventions: Other: AF screening

INTERVENTIONS:
Other: AF screening — Screening of AF in an opportunistic screening program using a smartphone device/application confirmed by ECG

SUMMARY:
Question: Can atrial fibrillation (AF) cases in patients ≥ 65 years be easily detected in a primary healthcare environment using a smartphone device and iECG application as an opportunistic screening tool?

Objectives:

Detection of AF through cardiac rhythm abnormalities in patients ≥65 years old in an opportunistic screening program using a smartphone device/application

1. Define the predictable value of the smartphone device with electrocardiogram (ECG) confirmation to detect AF in patients 65 years and older
2. Correlate screened patients cardiovascular risk profile and those that register cardiac rhythm irregularities for a better description of the general characteristics of Colombian population

ELIGIBILITY:
Inclusion Criteria:

* Females and males patients ≥65 years old attending primary care counselling
* Written informed consent

Exclusion Criteria:

* Patients with confirmed diagnosis of AF
* Patients who do not want to participate
* Patients consulting for acute conditions
* Patients presenting any diagnosed arrhythmia different than AF

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Subjects included in the study are patients 65 years and older reaching programmed primary care counselling, and who are willingly to participate and do not present any exclusion criteria for the screening
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients screened in whom the screening device detect an abnormal cardiac rhythm | Up to 6 months
Number of patients screened in whom Atrial Fibrillation (AF) was confirmed with ECG | Up to 6 months

SECONDARY OUTCOMES:
Number of patients in whom abnormal cardiac rhythm was detected with screening device and AF was confirmed with ECG | Up to 6 months
  Predictive value tests - Positive: Number of patients screened in whom AF was confirmed with ECG/ Number of patients screened in whom the screening device detect an abnormal rhythm - Negative: Number of patients screened in whom AF was discarded with ECG/ Number of patients screened in whom the screening device detect an abnormal rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer